CLINICAL TRIAL: NCT04880447
Title: Special Investigation of COMIRNATY Intramuscular Injection (Investigation of Patients With Underlying Disease Considered to be at High Risk of Aggravation of COVID-19)
Brief Title: Special Investigation of COMIRNATY in the Population With Underlying Diseases
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591019
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-01

CONDITIONS: COVID-19
Keywords: COVID-19,; Post-Marketing study; COMIRNATY; Underlying Disease
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COMIRNATY: COVID-19 mRNA vaccine
  Interventions: Biological: BNT162b2

INTERVENTIONS:
Biological: BNT162b2 — COMIRNATY is administered intramuscularly after dilution as a course of 2 doses (0.3 mL each). It is recommended to administer the second dose 3 weeks after the first dose.
  Other Names: COMIRNATY

SUMMARY:
Post-marketing study, Cohort study of COMIRNATY vaccines. To collect information on adverse events and COVID-19 observed after vaccination with COMIRNATY and to assess safety in patients with underlying disease considered to be at high risk of aggravation of COVID-19 who have received vaccination with this product under actual use conditions.

DETAILED DESCRIPTION:
This is a multicenter cohort study to be conducted in individuals with underlying diseases considered to be at high risk of aggravation of COVID-19 who are vaccinated with this product, and the investigator will enter the information required in this study in the case report forms (CRFs) based on the information obtained through preliminary examination sheet or medical interview, etc. and records such as medical records. A health observation diary will be distributed to the subjects participating in this study and they will be requested to record information on local reactions and systemic reactions after vaccination with this product.

ELIGIBILITY:
Inclusion Criteria:

-Subjects who are able to understand the content of this study and to record their symptoms in the health observation diary, and who have provided written consent to participate in this survey by themselves (or parents or legal guardians in the case of minors)

Exclusion Criteria:

* There are no exclusion criteria for this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with underlying disease considered to be at high risk of aggravation of COVID-19 (Underlying diseases considered to be at high risk of aggravation of COVID-19 are based on the range of patients with underlying diseases indicated by the Ministry of Health, Labour and Welfare for priority vaccination.)
Sampling Method: Probability Sample
Enrollment: 1075 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Local County, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591019

RESULTS

PARTICIPANT FLOW:
Groups:
- COMIRNATY Intramuscular Injection (Tozinameran): Participants with underlying disease considered to be at high risk of aggravation of COVID-19, who were vaccinated with Comirnaty as indicated in the approved local product document were observed from the date of Dose 1 to 28 days after Dose 2.
Period: Overall Study
Arm/Group | COMIRNATY Intramuscular Injection (Tozinameran)
Started | 1075
Completed | 1038
Not Completed | 37
Not completed — No vaccination information | 1
Not completed — No adverse event information (missing information) | 1
Not completed — Disease not covered in this study | 35

BASELINE CHARACTERISTICS:
Population: A total of 1075 participants were enrolled in this study. Of the 1075 participants from whom CRFs were collected, 37 participants were excluded from the safety analysis set due to the following reasons: No vaccination information (1 participant), No adverse event information (missing information) (1 participant), Disease not covered in this study (35 participants).
Arm/Group | COMIRNATY Intramuscular Injection (Tozinameran)
Number analyzed (Participants) | 1038
Age, Customized [Number; unit: Participants]
  <15 years | 3
  ≥15 and <65 years | 568
  ≥65 years | 467
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 433
  Male | 605
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Adverse Reactions
Description: An adverse reaction was any untoward medical occurrence attributed to COMIRNATY in a participant who was vaccinated with COMIRNATY. Relatedness to COMIRNATY was assessed by the physician. The proportion of adverse reactions was presented for the overall observation period, the observation period from the date of the first dose of Comirnaty up to 28 days after the second dose, and the observation period from the date of Dose 1 up to 28 days after Dose 2.
Time Frame: From the date of the first dose to 28 days after the second dose, up to approximately 49 days.
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and were vaccinated with COMIRNATY at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | COMIRNATY Intramuscular Injection (Tozinameran)
Number analyzed (Participants) | 1038
Participants
  Overall observation period | 59
  Observation from the 1st to the 2nd vaccination | 30
  Observation from 2nd vaccination to 28 days: number analyzed (Participants) | 1032
  Observation from 2nd vaccination to 28 days | 39

2. Primary Outcome: Proportion of Participants With Serious Adverse Reactions
Description: A serious adverse reaction was any untoward medical occurrence attributed to COMIRNATY resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; or congenital anomaly. Relatedness to COMIRNATY was assessed by the physician. The proportion of serious adverse reactions was presented for the overall observation period, the observation period from the first to the second vaccination, and the observation period from the date of Dose 1 up to 28 days after Dose 2.
Time Frame: From the date of the first dose to 28 days after the second dose, up to approximately 49 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | COMIRNATY Intramuscular Injection (Tozinameran)
Number analyzed (Participants) | 1038
Participants
  Overall observation period | 3
  Observation from the 1st to the 2nd vaccination | 1
  Observation from 2nd vaccination to 28 days: number analyzed (Participants) | 1032
  Observation from 2nd vaccination to 28 days | 2

3. Primary Outcome: Proportion of Participants With Local Reactions and Systemic Reactions (The First Vaccination)
Description: Local and systemic reactions were treated as specific adverse events of interest in this study, and were reported using the health observation diary filled out by the participants. Severity was rated and recorded as grade 1, 2, or 3 according to the FDA Guidance for industry: toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials. Health observation diary for the first vaccination was collected from 1035 participants of the 1038 safety analysis set participants.
Time Frame: Within 8 days after the date of the first dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- COMIRNATY Intramuscular Injection (Tozinameran) First COMIRNATY Vaccination Total (≥Grade 1): Participants with underlying disease considered to be at high risk of aggravation of COVID-19, who were vaccinated with Comirnaty as indicated in the approved local product document were observed within 8 days after Dose 1.
Arm/Group | COMIRNATY Intramuscular Injection (Tozinameran) First COMIRNATY Vaccination Total (≥Grade 1)
Number analyzed (Participants) | 1035
Participants
  Local reactions | 836
  Systemic reactions | 648

4. Primary Outcome: Proportion of Participants With Local Reactions and Systemic Reactions (The Second Vaccination)
Description: Local and systemic reactions were treated as specific adverse events of interest in this study, and were reported using the health observation diary filled out by the participants. Severity was rated and recorded as grade 1, 2, or 3 according to the FDA Guidance for industry: toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials. Health observation diary for the second vaccination was collected from 1026 participants of the 1032 participants who received the second vaccination with Comirnaty.
Time Frame: Within 8 days after the date of the second dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- COMIRNATY Intramuscular Injection (Tozinameran) Second COMIRNATY Vaccination Total (≥Grade 1): Participants with underlying disease considered to be at high risk of aggravation of COVID-19, who were vaccinated with Comirnaty as indicated in the approved local product document were observed within 8 days after Dose 2.
Arm/Group | COMIRNATY Intramuscular Injection (Tozinameran) Second COMIRNATY Vaccination Total (≥Grade 1)
Number analyzed (Participants) | 1026
Participants
  Local reactions | 866
  Systemic reactions | 716

ADVERSE EVENTS:
Time Frame: From the date of the first dose to 28 days after the second dose, up to approximately 49 days.
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | COMIRNATY Intramuscular Injection (Tozinameran)
All-Cause Mortality (participants affected / at risk) | 1/1038
Serious Adverse Events (participants affected / at risk) | 11/1038
Other Adverse Events (participants affected / at risk) | 114/1038
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | COMIRNATY Intramuscular Injection (Tozinameran) (N=1038)
Angina unstable (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Bacteraemia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Brain stem haemorrhage (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Intraventricular haemorrhage (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | COMIRNATY Intramuscular Injection (Tozinameran) (N=1038)
Anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Conjunctivitis allergic (Eye disorders) | 2
Ocular hyperaemia (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Faeces soft (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Paraesthesia oral (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Axillary pain (General disorders) | 2
Injection site bruising (General disorders) | 2
Injection site paraesthesia (General disorders) | 1
Injection site pruritus (General disorders) | 2
Malaise (General disorders) | 2
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 2
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 2
Thirst (General disorders) | 1
Vaccination site pruritus (General disorders) | 4
Vaccination site rash (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Abscess limb (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 2
Cystitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 5
Otitis externa (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1
Muscle injury (Injury, poisoning and procedural complications) | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1
Blood pressure decreased (Investigations) | 1
Blood pressure increased (Investigations) | 2
Brain natriuretic peptide increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Carpal tunnel syndrome (Nervous system disorders) | 1
Cervicobrachial syndrome (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Loss of consciousness (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 3
Taste disorder (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Chronic eosinophilic rhinosinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT04880447/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT04880447/SAP_001.pdf